CLINICAL TRIAL: NCT00568230
Title: An Open-Label, Single-Arm Feasibility Study of the Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty (PTMA) Device Used to Reduce Mitral Regurgitation.
Brief Title: Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty Device to Reduce Mitral Regurgitation
Acronym: PTOLEMY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viacor (Industry)
Responsible Party: Katharine M Stohlman, Viacor, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-023P
Record Dates: First submitted 2007-11-30; First posted 2007-12-05 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Heart Failure; Mitral Regurgitation
Keywords: heart failure; mitral regurgitation
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patient is screened for study, and given baseline assessments. Patient receives a diagnostic PTMA assessment and if responsive, receives a PTMA implant.
  Interventions: Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant

INTERVENTIONS:
Device: PTMA (Percutaneous Transvenous Mitral Annuloplasty) Implant — Percutaneous access from right or left subclavian vein with placement of assessment and placement of PTMA Implant into the coronary sinus, great cardiac vein. Device remains accessible from a subclavicular pocket.

SUMMARY:
Improvement of heart failure with moderate to severe mitral regurgitation using a percutaneously delivered implanted device.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic heart failure
* moderate to severe mitral regurgitation
* 20 - 50% LVEF

Exclusion Criteria:

* mitral regurgitation of organic origins
* recent interventions
* severe comorbidities

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
percent of patients who remain free from device-related major adverse events (death, myocardial infarction, tamponade, emergent cardiac surgery) | 30 days

SECONDARY OUTCOMES:
percent of implanted patients who maintain a sustained 1 grade reduction in mitral regurgitation and reduction of mitral annulus anterior posterior dimension | 30 days
improvement of clinical symptoms of heart failure as defined by percent of patients who exhibit one of the following: decrease in NYHA class, improvement in Minnesota QOL survey, increase in exercise capacity: 6 minute walk or VO2max | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sack, MD, Principal Investigator — Universitat Duisburg-Essen
Locations (1):
- Universitat Duisburg-Essen, Essen, Germany